CLINICAL TRIAL: NCT06819163
Title: Evaluation of the Effects of Berry Leaf Extract on Cognitive Processing in Healthy Elderly Adults
Acronym: SLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seppic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SLE
Record Dates: First submitted 2025-01-28; First posted 2025-02-11 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Cognitive Performance
Keywords: Memory; Attention; Stress; Elderly; Berry leaf extract

STUDY DESIGN:
Intervention Model Description: Comparative, randomized, placebo-controlled, double-blind, monocentric interventional study in parallel groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Berry leaf extract (Experimental): Dietary supplement - Berry leaf extract
  Interventions: Dietary Supplement: Berry leaf extract
- Placebo (Placebo Comparator): Dietary supplement - Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Berry leaf extract — The study foresees the intake of 2 capsules per day during 12 weeks
  Arms: Berry leaf extract
Dietary Supplement: Placebo — The study foresees the intake of 2 capsules per day during 12 weeks
  Arms: Placebo

SUMMARY:
This study aims to explore the positive effect of a dietary supplement composed of berry leaf extract on the cognitive performance and regulation of stress, mood, sleep and fatigue in healthy elderly adults with self-reported memory complaints

DETAILED DESCRIPTION:
This study is designed as a randomized double-blind placebo-controlled interventional study. One hundred and six participants (aged between 60 and 80), with self-perceived memory complaints, will be randomly allocated to the control (placebo supplement) or test (active supplement) group. Participants will be supplemented during 12 weeks with those products. Cognitive performance and psychological and emotional processing will be measured with tests and questionnaires before (baseline), at the middle (6 weeks), and at the end (12 weeks) of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Healthy woman or man
* Aged of 60 to 80 years (inclusive)
* With self-perceived memory complaints (CDS score ≥ 15)
* With a Body Mass Index (BMI) comprised between 18 and 30 kg/m2 (included)
* Participants must have completed a minimum of 12 years of formal education, starting from the age of 6. This corresponds to an education level equivalent to the completion of secondary school (e.g., a high school diploma or equivalent)
* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Stated willingness to maintain their usual life habits (diet, physical activity, alcohol consumption…)
* Speaking French

Exclusion Criteria:

* Subject with severe medical or cognitive problems which, in the opinion of the Principal Investigator, could interfere with the evaluation of the study criteria or with participant safety
* Subject with a MMSE score ≤ 24
* Subject with a coffee consumption of more than 5 cups per day
* Subject consuming drugs and/or with historical drug addiction (<5 years)
* Subject with a regular alcohol consumption exceeding 3 standard drinks per day (10 g of pure alcohol each), equivalent to 3 glasses of wine (12 cl), 3 glasses of beer (5°, 25cl), or 3 glasses of spirits (18°, 7 cl)
* Smoker or subject consuming regularly products containing nicotine
* Subject following a vegetarian or vegan diet
* Subject with known hypersensitivity to any component of the study product
* Subject who has taken in the 28 days preceding the screening visit or is currently taking drugs or food supplements aiming at improving memory, concentration, sleep, stress, anxiety or other substances which could, in the opinion of the Principal Investigator, interfere with cognitive and emotional processing
* Subject participating in another intervention trial

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Change in spatial working memory performance | 6 and 12 weeks
  Comparison between groups of the adjusted for baseline spatial working memory performance (number of errors) assessed by the Spatial Working Memory (SWM) subtest of the Cambridge Neuropsychological Test Automated Battery (CANTAB).

SECONDARY OUTCOMES:
Change in attentional performance | 6 and 12 weeks
  Comparison between groups of the adjusted for baseline attentional performance (reaction time) assessed by the Motor Screening Task subtest of the Cambridge Neuropsychological Test Automated Battery (CANTAB).
Change in psychomotor speed | 6 and 12 weeks
  Comparison between groups of the adjusted for baseline psychomotor speed (reaction time) assessed by the Reaction Time (RTI) subtest of the Cambridge Neuropsychological Test Automated Battery (CANTAB).
Change in verbal memory performance | 6 and 12 weeks
  Comparison between groups of the adjusted for baseline verbal memory performance (number of words, number of correct and incorrect responses) assessed by the Verbal Recognition Memory (VRM) subtest of the Cambridge Neuropsychological Test Automated Battery (CANTAB).
Change in visual memory performance | 6 and 12 weeks
  Comparison between groups of the adjusted for baseline visual memory performance (number or errors, number of trials and number of stages completed) assessed by the Paired Associates Learning (PAL) subtest of the Cambridge Neuropsychological Test Automated Battery (CANTAB).
Change in executive functions' performance | 6 and 12 weeks
  Comparison between groups of the adjusted for baseline executive functions performance (number of errors) assessed by the Multitasking Test (MTT) subtest of the Cambridge Neuropsychological Test Automated Battery (CANTAB).
Evolution of self-perceived emotional status | 6 and 12 weeks
  Comparison between groups of the adjusted for baseline self-perceived level of emotions assessed by the Positive and Negative Affect Schedule (PANAS) questionnaire. Items are rated on a scale ranging from 1 = very slightly or not at all to 5 = extremely.
Evolution of sleep quality | 6 and 12 weeks
  Comparison between groups of the adjusted for baseline sleep quality assessed by the Insomnia Severity Index (ISI) questionnaire. Items are rated on a scale ranging from 0 = no problem to 4 = very severe problem.
Evolution of self-perceived level of stress | 6 and 12 weeks
  Comparison between groups of the adjusted for baseline of self-perceived level of stress assessed by the Perceived Stress Scale (PSS-10) questionnaire. Items are rated on a scale ranging from 0 = never to 4 = very often.
Evolution of fatigue level | 6 and 12 weeks
  Comparison between groups of the adjusted for baseline of level of fatigue assessed by the Fatigue Assessment Scale (FAS) questionnaire. Items are rated on a scale ranging from from 1 = never to 5 = always.
Evolution of self-perceived cognitive difficulties | 6 and 12 weeks
  Comparison between groups of the adjusted for baseline of self-perceived cognitive difficulties assessed by the Cognitive Difficulties Scale (CDS) questionnaire. Items are rated on a scale ranging from 0 = never to 3 = most of the time.
Evolution of self-rated general subjective health | 6 and 12 weeks
  Comparison between groups of the adjusted for baseline of self-rated general subjective health assessed by a visual analogue scale, ranging from 1 = very bad to 5 = very good.
Evolution of self-perceived enhancement of memory | 6 and 12 weeks
  Comparison between groups of the adjusted for baseline of self-perceived enhancement of memory by a visual analogue scale, ranging from 0 = not at all to 4 = very much.
Evolution of self-perceived enhancement of concentration | 6 and 12 weeks
  Comparison between groups of the adjusted for baseline of self-perceived enhancement of concentration assessed by a visual analogue scale, ranging from 0 = not at all to 4 = very much.
Evolution of self-perceived enhancement of attention | 6 and 12 weeks
  Comparison between groups of the adjusted for baseline of self-perceived enhancement of attention assessed by a visual analogue scale, ranging from 0 = not at all to 4 = very much.

CONTACTS AND LOCATIONS:
Overall Officials: Louise Deldicque, Pr, Study Director — Université Catholique de Louvain; Sylvie Copine, Dr, Principal Investigator — Université Catholique de Louvain; Laurent Simar, Dr, Principal Investigator — Université Catholique de Louvain
Locations (1):
- Center of Investigation in Clinical Nutrition (CICN), Louvain-la-Neuve, Belgium

IPD SHARING:
Plan to Share IPD: No